CLINICAL TRIAL: NCT07022626
Title: A Randomised Controlled Trial Assessing the Value of Computed Tomography Cardiac Angiography in Improving Patient Satisfaction and Reducing Contrast Load, Procedural Duration and Complications in Patients Who Had Previous Bypass Surgery Undergoing Coronary Angiography
Brief Title: Trial to Assess Whether Computed Tomography Cardiac Angiography Can Improve Invasive Coronary Angiography in Bypass Surgery Patients
Acronym: BYPASS-CTCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Reda 012466
Record Dates: First submitted 2024-11-04; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Ischaemic Heart Disease; Contrast-induced Nephropathy
Keywords: Coronary Artery Bypass Grafts; Computed Tomography Coronary Angiography; Invasive Coronary Angiogram
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTCA + ICA (Active Comparator): Computed Tomography Cardiac Angiography (CTCA) performed prior to invasive coronary angiography (ICA).
  Interventions: Procedure: CTCA
- ICA only (No Intervention): Invasive coronary angiography (ICA) performed only.

INTERVENTIONS:
Procedure: CTCA — Computed Tomography Coronary Angiography (CTCA) performed prior to invasive coronary angiography (ICA)
  Other Names: Computed Tomography Coronary Angiogram
  Arms: CTCA + ICA

SUMMARY:
A large number of patients with symptomatic ischaemic heart disease undergo coronary artery bypass grafting (CABG) to alleviate their symptoms and improve prognosis. Given the progressive nature of coronary disease, bypass grafts can narrow or block over time, leading to chest pain and the need for further invasive coronary angiography. Invasive coronary procedures in patients with bypass grafts can be more complicated due to the variation in bypass graft ostia. This can lead to longer procedure times, with higher doses of contrast and radiation and more discomfort for the patient. The aim of this study is to see if the use of computed tomography coronary angiography (CTCA) in patients with previous bypass grafts prior to invasive coronary angiography will help make their procedure safer and quicker.

DETAILED DESCRIPTION:
The BYPASS-CTCA trial is a single-centre, randomised controlled trial, which plans to recruit 688 patients who have had previous bypass grafts and require invasive coronary angiography over a period of 30 months.

Patients will be randomised to receive either computed tomography coronary angiography (CTCA) prior to their invasive coronary angiogram, or invasive coronary angiography alone.

The primary endpoints will be the incidence of contrast induced nephropathy, the duration of the invasive coronary angiographic procedure and patient satisfaction. A number of secondary endpoints will also be looked at.

Findings from BYPASS-CTCA will potentially demonstrate that a CTCA prior to invasive coronary angiography in this cohort of patients reduces the incidence of contrast-induced kidney injury, the length of procedure and improves patients satisfaction. The results of this trial may influence future clinical practice guidelines in coronary artery bypass graft patients undergoing invasive coronary procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing coronary angiography +/-Percutaneous coronary Intervention
2. Previous Coronary Artery Bypass Grafting (CABG)
3. Aged ≥18
4. Patients able and willing to give their written informed consent.

Exclusion Criteria:

1. Subjects presenting with ST elevation myocardial infarction, cardiogenic shock (systolic blood pressure <80 mmHg for >30 minutes, or requiring inotropes or emergency intra aortic balloon pump for hypotension treatment) or cardiopulmonary resuscitation.
2. Subjects with eGFR <20ml/min or on renal replacement therapy.
3. Current life-threatening condition other than vascular disease that may prevent a subject completing the study.
4. Clinical instability including cardiogenic shock, hypotension (low blood pressure-systolic blood pressure less than 90 mmHg), sustained ventricular or atrial arrhythmia requiring intravenous medications.
5. Inability to tolerate beta-blockers, including those with chronic obstructive pulmonary disease or asthma, complete heart block, second-degree atrioventricular block
6. Known contrast dye allergy.
7. Pregnancy or unknown pregnancy status.
8. Patients considered unsuitable to participate by the research team (e.g., due to medical reasons, laboratory abnormalities, or subject's unwillingness to comply with all study related procedures).
9. Inability or refusal to provide informed consent.
10. Any inclusion criteria not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Procedural duration | timer started after the insertion of the arterial catheter and stopped when the catheters are removed
  To measure the length of coronary angiographic procedure
Incidence of Contrast Induced Nephropathy | 48-72 hours
  Defined by Kidney Disease: Improving Global Outcomes (KDIGO) criteria
Patient Satisfaction | 4-6 hours post angiogram +/- percutaneous coronary intervention
  Patient satisfaction measured by validated questionnaire

SECONDARY OUTCOMES:
Contrast Amount | During procedure
  Contrast amount (mls) administered during invasive coronary angiography
Radiation Exposure | During procedure
  Radiation exposure (mSv) during invasive coronary angiography
Angiography Related Complications | During procedure
  Angiography related complications (such as coronary or aortic dissection, stroke, bleeding, vascular access complication)
Radial Access Rate | During procedure
  Radial access rates during invasive coronary angiography
Catheters Used | During procedure
  Number of catheters used during invasive coronary angiography
Computed Tomography Cardiac Angiography Accuracy | Computed Tomography Cardiac Angiography (CTCA)
  Accuracy of the computed tomography cardiac angiography scan for detecting graft patency
Number of grafts not identified | During procedure
  Number of grafts not identified during invasive coronary angiography
Cost effectiveness of computed tomography cardiac angiography | 12 months
  Cost effectiveness of the intervention (per quality-adjusted life years) measured over 12 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jones, MRCP, PhD, Principal Investigator — Queen Mary University of London
Locations (2):
- United Kingdom (2):
  - Royal London Hospital, London
  - St Bartholomew's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
The trial protocol will be published
Supporting Information: Study Protocol
Time Frame: Mid-late 2018
Access Criteria: Freely available via journal